CLINICAL TRIAL: NCT04570553
Title: Use of an Intrauterine Manipulator and Its Correlation with Positive Peritoneal Cytology in Early Stage Endometrial Cancers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: WellSpan Health (Other)
Responsible Party: Principal Investigator, Eav Lim, Site Director, Gynecology Oncology, WellSpan Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1627644
Record Dates: First submitted 2020-09-25; First posted 2020-09-30 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-04

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; peritoneal cytology
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: Subjects are randomized to one of two groups in parallel: V-care uterine manipulator group or sponge stick group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- V-care uterine manipulator (Experimental): Patients in the V-care uterine manipulator arm will undergo standard staging surgery utilizing a V-care uterine manipulator in the standard fashion
  Interventions: Procedure: surgical staging
- Sponge stick (Active Comparator): Patients in the sponge stick arm will undergo standard staging surgery utilizing a non-invasive sponge stick for cervical delineation.
  Interventions: Procedure: surgical staging

INTERVENTIONS:
Procedure: surgical staging — Patients will undergo standard surgical staging for endometrial cancer utilizing either a V-care uterine manipulator or sponge stick

SUMMARY:
This study aims to answer whether use of a Vcare® intrauterine manipulator leads to an increased incidence of positive peritoneal cytology in patients undergoing surgical management of early stage (FIGO stage I/II) endometrial cancer.

DETAILED DESCRIPTION:
Endometrial cancer is the sixth most common cancer diagnosed in women worldwide and the leading gynecologic cancer in developed countries, accounting for nearly 50% of all newly diagnosed gynecologic cancers in the United States . The majority of endometrial cancers are diagnosed at an early stage which portends a favorable prognosis. Despite early diagnosis and generally favorable prognosis in these cancers, approximately 13% of patients will experience recurrence . Most recurrences occur in patients with known high-risk pathologic features, however approximately 3% of recurrences occur in patients with no high-risk pathology features . While well-defined pathologic factors such as age, tumor grade, and depth of invasion have been described for high-risk of recurrence, predicting recurrence in low-risk patients has been an ongoing challenge in the management of early stage endometrial cancers

One potential contribution to recurrence in low-risk endometrial cancers may be the presence of positively malignant peritoneal cytology. Positive peritoneal cytology (PPC) has been an ongoing topic of debate regarding its significance and optimal management in early stage endometrial cancers. Creasman and Rutledge initially described the prognostic value of peritoneal cytology in 1971 by linking PPC with worse survival at 4 years . Since then multiple studies have sought to address the significance of peritoneal cytology in endometrial cancer, many with conflicting results. Studies by Kasamatsu et al, Fadare et al, Lurain et al and Scott et al found that PPC is not a significant prognostic factor for disease recurrence or survival . Contrary to these data however studies by Lee et al, Garg et al, and Seagle et al have shown a positive correlation with PPC as both a prognostic factor and survival . Despite these conflicting data directing the significance of PPC, it remains an important contributing factor in the management and prognosis of endometrial cancer. Although peritoneal cytology was removed from FIGO staging in 2009, NCCN guidelines continue to recommend the collection of peritoneal cytology in order to further elucidate the impact of PPC, with some authors calling for the reinstatement of peritoneal cytology in endometrial cancer staging .

In addition to the effects of pathological factors and peritoneal cytology on recurrence risk, recent studies in other gynecologic cancers have shown how different approaches in surgical management play a key role in overall disease prognosis and outcomes. The LACC trial, published in 2018, demonstrated the effects of differing surgical technique on outcomes by showing that patients undergoing minimally invasive surgery for management of cervical cancers fared worse in locoregional recurrence, disease-free survival and overall survival than patients undergoing traditional laparotomy. This study highlights the impact of surgical methodology on the prognosis and outcomes of oncologic surgery.

Similar to the management of cervical cancers, over the last two decades laparoscopic surgery and staging has become the mainstay of management for women with uterine cancers. The traditional approach of laparotomy with hysterectomy, bilateral salpingo-oophorectomy, pelvic and para-aortic lymphadenectomy has come to be effectively replaced with the minimally invasive, laparoscopic approach which affords an equally efficacious surgery with shorter recovery and fewer complications . In order to perform more efficient and safe surgeries, intrauterine manipulators have been employed in laparoscopic hysterectomy. Since their introduction into gynecologic oncology surgery questions have risen regarding the possibility of increased risk of tumor dissemination with usage of intrauterine manipulators. The mechanisms of this have been theorized to include retrograde dissemination via the fallopian tubes into the peritoneal cavity as well as increased lymphovascular space invasion . Multiple studies have focused on the question of retrograde dissemination via the fallopian tubes with conflicting results. A retrospective study by Sonoda et el found that when low-risk endometrial cancer was managed with laparoscopic assisted vaginal hysterectomy (LAVH) using an inflatable intrauterine manipulator, it was associated with increased incidence of positive peritoneal cytology compared to the control population (10.3% versus 2.8%). Lim et al prospectively evaluated the effect of uterine manipulator use on peritoneal cytology in laparoscopic hysterectomy using a RUMI manipulator and KOH colpotomizer and found that 4.3% of patients in their study were upstaged due to PPC following usage of a uterine manipulator . However, contrary to this, two prospective studies found that usage of a uterine manipulator did not increase the incidence of malignant peritoneal cytology in patients undergoing laparoscopic staging. A prospective study by Eltabakh et al evaluated conversion from negative to PPC immediately following insertion of a Pelosi uterine manipulator in 42 patients. Based on their results that demonstrated no patients converted to PPC, they concluded that intrauterine manipulators do not increase the incidence of PPC. Additionally, Lee et al published results of a randomized parallel trial of 110 patients undergoing laparoscopic surgery and staging for stage I endometrial cancer either with or without a uterine manipulator which showed no significant difference in the rate of positive cytology in either group.

This study will be a randomized control trial in which patients will be randomized into two study arms following informed consent: a control arm utilizing a non-invasive sponge stick (Foerster ring forceps containing a raytec sponge (Vistec Covidien Health, Mansfield, MA)) placed in the vagina for surgical assistance or a Vcare® intrauterine manipulator (ConMed Endosurgery, Utica, NY). Patients randomized to the Vcare® group will have the Vcare® placed in the usual fashion under direct visualization following entrance into the abdomen. Cytology washings will be obtained following entrance into the peritoneal cavity. Washings will be obtained by washing approximately 150cc of normal saline over the bilateral paracolic gutters, uterine fundus, and anterior and posterior cul de sacs. Fifty milliliters of fluid will then be aspirated for cytology collection. Cytology washings will then be obtained again prior to colpotomy. Patients will undergo total laparoscopic hysterectomy or robotic assisted total laparoscopic hysterectomy. Peritoneal washings obtained during surgery will be processed and undergo pathological examination. Covariate data including age, BMI, history of previous tubal ligation, FIGO stage, histologic type, histologic grade, lymphovascular space invasion, and gross evidence of tumor spillage will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 18 or older able to give informed consent
* Biopsy diagnosed endometrial cancer (including endometrioid, serous, mucinous and clear cell histologies)
* Planned standard of care surgical management of early stage endometrial cancer
* No clinical evidence of disseminated intraperitoneal disease

Exclusion Criteria:

* Final pathology does not reflect diagnosis of endometrial cancer (including endometrioid, serous, mucinous, and clear cell histology)
* Evidence of disseminated intraperitoneal disease
* Subject is not a surgical candidate
* Subject elects for fertility sparing or non-operative management
* Subject is unable to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female subjects age 18 and older
Enrollment: 350 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Conversion of positive peritoneal cytology | 2 years
  Intraoperative conversion rate from negative to positive peritoneal cytology will be assessed in each arm

SECONDARY OUTCOMES:
Recurrence rate | 2 years
  Endometrial cancer rates at 2 years from surgery will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Eav Lim, DO, Principal Investigator — WellSpan Health
Locations (1):
- Wellspan Health, York, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Cancer Research Fund/American Institute for Cancer Research. Diet, Nutrition, Physical Activity and Cancer: a Global Perspective. Continuous Update Project Expert Report 2018. Available at dietandcancerreport.org.
- [Background] Campos SM, Lee LJ, Del Carmen, MG, McMeekin DS. Corpus: Epithelial Tumors. In DS Chi, A Berchuk, DS Dizon, and CM Yashar (Eds.), Principles and Practice of Gynecologic Oncology. (pp 511) Philadelphia, PA: Wolters Kluwer.
- [Background] Fung-Kee-Fung M, Dodge J, Elit L, Lukka H, Chambers A, Oliver T; Cancer Care Ontario Program in Evidence-based Care Gynecology Cancer Disease Site Group. Follow-up after primary therapy for endometrial cancer: a systematic review. Gynecol Oncol. 2006 Jun;101(3):520-9. doi: 10.1016/j.ygyno.2006.02.011. Epub 2006 Mar 23. PMID 16556457
- [Background] Creasman WT, Morrow CP, Bundy BN, Homesley HD, Graham JE, Heller PB. Surgical pathologic spread patterns of endometrial cancer. A Gynecologic Oncology Group Study. Cancer. 1987 Oct 15;60(8 Suppl):2035-41. doi: 10.1002/1097-0142(19901015)60:8+3.0.co;2-8. PMID 3652025
- [Background] Creutzberg CL, van Putten WL, Koper PC, Lybeert ML, Jobsen JJ, Warlam-Rodenhuis CC, De Winter KA, Lutgens LC, van den Bergh AC, van de Steen-Banasik E, Beerman H, van Lent M. Surgery and postoperative radiotherapy versus surgery alone for patients with stage-1 endometrial carcinoma: multicentre randomised trial. PORTEC Study Group. Post Operative Radiation Therapy in Endometrial Carcinoma. Lancet. 2000 Apr 22;355(9213):1404-11. doi: 10.1016/s0140-6736(00)02139-5. PMID 10791524
- [Background] Creasman WT, Rutledge F. The prognostic value of peritoneal cytology in gynecologic malignant disease. Am J Obstet Gynecol. 1971 Jul 15;110(6):773-81. doi: 10.1016/0002-9378(71)90571-0. No abstract available. PMID 5561996
- [Background] Kasamatsu T, Onda T, Katsumata N, Sawada M, Yamada T, Tsunematsu R, Ohmi K, Sasajima Y, Matsuno Y. Prognostic significance of positive peritoneal cytology in endometrial carcinoma confined to the uterus. Br J Cancer. 2003 Jan 27;88(2):245-50. doi: 10.1038/sj.bjc.6600698. PMID 12610496
- [Background] Fadare O, Mariappan MR, Hileeto D, Wang S, McAlpine JN, Rimm DL. Upstaging based solely on positive peritoneal washing does not affect outcome in endometrial cancer. Mod Pathol. 2005 May;18(5):673-80. doi: 10.1038/modpathol.3800342. PMID 15578078
- [Background] Lurain JR, Rumsey NK, Schink JC, Wallemark CB, Chmiel JS. Prognostic significance of positive peritoneal cytology in clinical stage I adenocarcinoma of the endometrium. Obstet Gynecol. 1989 Aug;74(2):175-9. PMID 2748053
- [Background] Scott SA, van der Zanden C, Cai E, McGahan CE, Kwon JS. Prognostic significance of peritoneal cytology in low-intermediate risk endometrial cancer. Gynecol Oncol. 2017 May;145(2):262-268. doi: 10.1016/j.ygyno.2017.03.011. Epub 2017 Mar 28. PMID 28359690
- [Background] Lee B, Suh DH, Kim K, No JH, Kim YB. Influence of positive peritoneal cytology on prognostic factors and survival in early-stage endometrial cancer: a systematic review and meta-analysis. Jpn J Clin Oncol. 2016 Aug;46(8):711-7. doi: 10.1093/jjco/hyw063. Epub 2016 May 20. PMID 27207885
- [Background] Garg G, Gao F, Wright JD, Hagemann AR, Mutch DG, Powell MA. Positive peritoneal cytology is an independent risk-factor in early stage endometrial cancer. Gynecol Oncol. 2013 Jan;128(1):77-82. doi: 10.1016/j.ygyno.2012.09.026. Epub 2012 Sep 29. PMID 23032094
- [Background] Seagle BL, Alexander AL, Lantsman T, Shahabi S. Prognosis and treatment of positive peritoneal cytology in early endometrial cancer: matched cohort analyses from the National Cancer Database. Am J Obstet Gynecol. 2018 Mar;218(3):329.e1-329.e15. doi: 10.1016/j.ajog.2017.11.601. Epub 2017 Dec 6. PMID 29223598
- [Background] Ramirez PT, Frumovitz M, Pareja R, Lopez A, Vieira M, Ribeiro R, Buda A, Yan X, Shuzhong Y, Chetty N, Isla D, Tamura M, Zhu T, Robledo KP, Gebski V, Asher R, Behan V, Nicklin JL, Coleman RL, Obermair A. Minimally Invasive versus Abdominal Radical Hysterectomy for Cervical Cancer. N Engl J Med. 2018 Nov 15;379(20):1895-1904. doi: 10.1056/NEJMoa1806395. Epub 2018 Oct 31. PMID 30380365
- [Background] Walker JL, Piedmonte MR, Spirtos NM, Eisenkop SM, Schlaerth JB, Mannel RS, Spiegel G, Barakat R, Pearl ML, Sharma SK. Laparoscopy compared with laparotomy for comprehensive surgical staging of uterine cancer: Gynecologic Oncology Group Study LAP2. J Clin Oncol. 2009 Nov 10;27(32):5331-6. doi: 10.1200/JCO.2009.22.3248. Epub 2009 Oct 5. PMID 19805679
- [Background] Walker JL, Piedmonte MR, Spirtos NM, Eisenkop SM, Schlaerth JB, Mannel RS, Barakat R, Pearl ML, Sharma SK. Recurrence and survival after random assignment to laparoscopy versus laparotomy for comprehensive surgical staging of uterine cancer: Gynecologic Oncology Group LAP2 Study. J Clin Oncol. 2012 Mar 1;30(7):695-700. doi: 10.1200/JCO.2011.38.8645. Epub 2012 Jan 30. PMID 22291074
- [Background] Logani S, Herdman AV, Little JV, Moller KA. Vascular "pseudo invasion" in laparoscopic hysterectomy specimens: a diagnostic pitfall. Am J Surg Pathol. 2008 Apr;32(4):560-5. doi: 10.1097/PAS.0b013e31816098f0. PMID 18300797
- [Background] Zhang C, Havrilesky LJ, Broadwater G, Di Santo N, Ehrisman JA, Lee PS, Berchuck A, Alvarez Secord A, Bean S, Bentley RC, Valea FA. Relationship between minimally invasive hysterectomy, pelvic cytology, and lymph vascular space invasion: a single institution study of 458 patients. Gynecol Oncol. 2014 May;133(2):211-5. doi: 10.1016/j.ygyno.2014.02.025. Epub 2014 Feb 28. PMID 24582867
- [Background] Sonoda Y, Zerbe M, Smith A, Lin O, Barakat RR, Hoskins WJ. High incidence of positive peritoneal cytology in low-risk endometrial cancer treated by laparoscopically assisted vaginal hysterectomy. Gynecol Oncol. 2001 Mar;80(3):378-82. doi: 10.1006/gyno.2000.6079. PMID 11263935
- [Background] Lim S, Kim HS, Lee KB, Yoo CW, Park SY, Seo SS. Does the use of a uterine manipulator with an intrauterine balloon in total laparoscopic hysterectomy facilitate tumor cell spillage into the peritoneal cavity in patients with endometrial cancer? Int J Gynecol Cancer. 2008 Sep-Oct;18(5):1145-9. doi: 10.1111/j.1525-1438.2007.01165.x. Epub 2008 Jan 22. PMID 18217979
- [Background] Eltabbakh GH, Mount SL. Laparoscopic surgery does not increase the positive peritoneal cytology among women with endometrial carcinoma. Gynecol Oncol. 2006 Feb;100(2):361-4. doi: 10.1016/j.ygyno.2005.08.040. Epub 2005 Sep 26. PMID 16185754
- [Background] Lee M, Kim YT, Kim SW, Kim S, Kim JH, Nam EJ. Effects of uterine manipulation on surgical outcomes in laparoscopic management of endometrial cancer: a prospective randomized clinical trial. Int J Gynecol Cancer. 2013 Feb;23(2):372-9. doi: 10.1097/IGC.0b013e3182788485. PMID 23266650